CLINICAL TRIAL: NCT02733055
Title: Posturography as Biomarker of Oculomotor and Postural Control Integration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CI-IRB-20160321002
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Postural Balance
Keywords: Postural Equilibrium; Musculoskeletal Equilibrium; Eye Movements; Saccades; Pursuit, Smooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subjects (Experimental): participant undergoing posturographic evaluation
  Interventions: Other: posturographic evaluation

INTERVENTIONS:
Other: posturographic evaluation — subjects will undergo CDP testing using one of the ext_mCTSIB tests without (baseline) and with oculomotor task

SUMMARY:
Determine the effects looking in certain direction or moving the eyes in a certain way have on the ability of a subject to maintain equilibrium in different circumstances (eyes open/closed, and standing on hard or compliant surface, with the head straight or rotated right or left, flexed or extended).

DETAILED DESCRIPTION:
Subjects will undergo computerized dynamic posturography (CDP) testing using the extended modified Clinical Testing of Sensory Integration in Balance (ext_mCTSIB) protocol: the subjects will be required to stand on a hard or the compliant surface in a comfortable posture, feet shoulder width, with eyes open or closed, arms to the side and free to move, gazing forward, and breathing normally, with head straight, turned right or left, flexed or extended. This testing will be used to determine the health status of the subjects.

Then a sequence of tests will be performed (they could be done in different days to avoid fatiguing the subject): each sequence will comprise of a baseline test in one of the ext_mCTSIB testing conditions and a subsequent test in the same conditions but with an oculomotor additional task, such as gazing in a specific direction other than straight, performing saccades in different directions, at different speed and using different paradigms (prosaccades, antisaccades, to a remembered target, gap saccades, …), following a target moving on the screen at different speed and in different directions, receiving an optokinetic stimulation in different directions and at different speeds. Video recordings of the eyes movement may be done to make sure that the subject is actually moving the eyes, to verify that the observers are well trained to detect and count the saccadic movements, as well as to obtain quantitative information regarding the eye movements per se.

ELIGIBILITY:
Inclusion Criteria:

* Self assessed healthy subjects

Exclusion Criteria:

* subjects suffering from pathology known to affect balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Stability Score | immediately after data collection
  The Stability Score (calculated as percentage ratio of the actual sway and the theoretical limit of stability) will be used to investigate if there is any difference between the test without and with oculomotor task. Statistical tools such t-tests and correlation coefficients will be used to assess if there is a difference between the two tests

SECONDARY OUTCOMES:
average velocity moment [mm^2/s] | immediately after data collection
  The average velocity moment (calculated as as the product of sway velocity path length) will be used to investigate if there is any difference between the test without and with oculomotor task. Statistical tools such t-tests and correlation coefficients will be used to assess if there is a difference between the two tests
sway path length [mm] | immediately after data collection
  The sway path length (the distance traveled during the test) will be used to investigate if there is any difference between the test without and with oculomotor task. Statistical tools such t-tests and correlation coefficients will be used to assess if there is a difference between the two tests
frequency content [Hz] | immediately after data collection
  The frequency content (calculated using FFT) will be used to investigate if there is any difference between the test without and with oculomotor task. Statistical tools such t-tests and correlation coefficients will be used to assess if there is a difference between the two tests

CONTACTS AND LOCATIONS:
Overall Officials: Paul Noone, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (2):
- Carrick Institute for Graduate Studies, Atlanta, Georgia, United States
- Carrick Institute for Graduate Studies, Hampton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No